CLINICAL TRIAL: NCT04763304
Title: Self-contamination Following Removal of Two Personal Protective Equipment Suits: a Randomized, Controlled, Crossover Simulation Trial
Brief Title: Self-contamination Following Removal of Two Personal Protective Equipment Suits: a Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, DELFINA SANCHEZ NOVAS, Physician, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 5646
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Personal Protective Equipment; Self Contamination
Keywords: sars-cov-2; personal protective equipment; self-contamination; fluorescent solution; healthcare simulation

STUDY DESIGN:
Intervention Model Description: We designed a prospective, randomized, controlled crossover trial with a total of 60 healthy anesthesia personnel volunteers. A two-period/two-intervention (AB/BA) design was chosen for this trial in order to estimate differences between both PPE suits with greater precision, given there is no participant variation between groups. The primary outcome was within-participant variability. A potential carryover effect was not expected considering the combination of an active (wet wipe cleansing) and passive (15 minute interval) washout period between interventions. All participants were randomly allocated to either intervention sequence: PPE-G (personal protective equipment including a gown for body protection) followed by PPE-C (personal protective equipment including a coverall for body protection) or PPE-C followed by PPE-G. Both interventions took place on the same day.
Who Masked: Outcomes Assessor
Masking Description: In a specific area, the blinded outcome assessor (researcher #2) performed standardized scanning of participants' skin and base clothing using ultraviolet light in a dark room, revealing the presence of any fluorescent traces. The seven body zones assessed were face, anterior and posterior neck, arms, hands, clothing (anterior/posterior, upper, and lower clothing), and foot covers. Fluorescent traces were measured (small traces, ≤1 cm; large traces, >1 cm) and quantified for statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPE-G (gown) followed by PPE-C (coverall) (Active Comparator): Placement of PPE-G (personal protective equipment including a gown for body protection) fluorescent solution full-body spray, removal of PPE-G and assessment of self-contamination through ultraviolet light scanning.
  Placement of PPE-C (personal protective equipment including a coverall for body protection), fluorescent solution full-body spray, removal of PPE-C and assessment of self-contamination through ultraviolet light scanning.
  Interventions: Other: Gown personal protective equipment (PPE-G) suit; Other: Coverall personal protective equipment (PPE-C) suit
- PPE-C (coverall) followed by PPE-G (gown) (Active Comparator): Placement of PPE-C (personal protective equipment including a coverall for body protection), fluorescent solution full-body spray, removal of PPE-C and assessment of self-contamination through ultraviolet light scanning.
  Placement of PPE-G (personal protective equipment including a gown for body protection), fluorescent solution full-body spray, removal of PPE-G and assessment of self-contamination through ultraviolet light scanning.
  Interventions: Other: Gown personal protective equipment (PPE-G) suit; Other: Coverall personal protective equipment (PPE-C) suit

INTERVENTIONS:
Other: Gown personal protective equipment (PPE-G) suit — Placement of PPE-G under direct instructions (audio recording), fluorescent solution full-body spray, removal of PPE under direct instructions (audio recording) and assessment of self-contamination through ultraviolet light scanning. Active (wet wipe cleanse of any fluorescent traces visible under ultraviolet light scanning) and passive (15 minute interval) washout period to prevent a carry over effect on the second allocated intervention.
Other: Coverall personal protective equipment (PPE-C) suit — Placement of PPE-C under direct instructions (audio recording), fluorescent solution full-body spray, removal of PPE under direct instructions (audio recording) and assessment of self-contamination through ultraviolet light scanning. Active (wet wipe cleanse of any fluorescent traces visible under ultraviolet light scanning) and passive (15 minute interval) washout period to prevent a carry over effect on the second allocated intervention.

SUMMARY:
Anesthesiologists and other professionals are at high risk of viral infection during aerosol-generating procedures. Knowledge of the protective quality of PPE suits and the risk of self-contamination after removal is paramount. This trial used an ultraviolet-fluorescent solution to explore differences in self-contamination after removal of gown PPE (PPE-G) and coverall PPE (PPE-C). A two-period/two-intervention (AB/BA) design was chosen; each intervention consisted of audio-guided placement of PPE, full-body spraying of fluorescent solution, audio-guided removal of PPE, and assessment of self-contamination through ultraviolet light scanning. The primary outcome was the mean within-participant difference (traces of any size) between PPE suits. Statistical significance was tested using t test for paired data.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology Department member (Hospital Italiano de Buenos Aires, Buenos Aires, Argentina), participation in the PPE training workshop.

Exclusion Criteria:

* Refusal to participate in the study
* Known allergy to any of the components of the fluorescent lotion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Mean within-participant difference in self-contamination between PPE-G and PPE-C suits | 20 minutes
  Mean difference between paired observations (number of fluorescent traces, any size, any body zone, per PPE suit) from each participant.

SECONDARY OUTCOMES:
Correlation between self-contamination and adherence to the PPE removal protocol | 5 minutes
  Graphical illustration of adherence in the "X" axis and number of traces in the "Y" axis and calculation of the Spearman's rank-order correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, ICF
Time Frame: At time of publication.